CLINICAL TRIAL: NCT05912582
Title: Prospective Study for Molecular Biomarkers and Spatial Transcriptomics of Nasopharyngeal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Lirong Wu, Associate Professor, Jiangsu Cancer Institute & Hospital
Other Study IDs: Biomarkers- NPC
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Biomarker; Spatial Transcriptomics
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood is obtained from patients when recruited, completing 10, 20, 32 fractions of radiation therapy, 3 months after radiation therapy and disease progression. Tumor tissue specimens are obtained from patients when recruited and disease progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation Group
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT) combined with chemotherapy

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy (IMRT) combined with chemotherapy — Intensity modulated radiation therapy (IMRT) combined with chemotherapy
  Other Names: IMRT

SUMMARY:
This clinical research aims to explore potential biomarkers and validate molecular signatures' predictive and prognostic value in nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Primary endpoint: Evaluation of the major pathological response of nasopharyngeal carcinoma patients.

Secondary endpoint: Evaluation of failure-free survival and overall survival of nasopharyngeal carcinoma patients.

Outline: This is a prospective observational study. Patients of nasopharyngeal carcinoma undergo inductive chemotherapy and concurrent chemoradiotherapy. Whole blood is obtained from patients when recruited, completing 10, 20, 32 fractions of radiation therapy, 3 months after radiation therapy and disease progression. Tumor tissue specimens are obtained from patients when recruited and disease progression. The samples are analyzed for biomarkers and spatial transcriptomics. The biomarkers and spatial transcriptomics are correlated with clinical outcomes (major pathological response, progression-free survival, overall survival, tumor response to treatment, distant metastasis, recurrence and death).

The analysis aims to explore potential biomarkers and validate molecular signatures' predictive and prognostic value in nasopharyngeal carcinoma. This will lead to the definition of risk groups and stratification of patients and will help in precision medicine of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed nasopharyngeal carcinoma
2. No evidence of distant metastasis (M0)
3. Written informed consent

Exclusion Criteria:

Treatment with palliative intent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly histologically confirmed stage IVa nasopharyngeal carcinoma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-06-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
major pathological response | 3 months after radiation therapy

SECONDARY OUTCOMES:
Progression-free Survival | 2 years after radiation therapy
Overall Survival | 2 years after radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol